CLINICAL TRIAL: NCT00985348
Title: Randomized, Monocenter, Open Label, Two-way Cross-over, Single Dose Bioequivalence Study of Two Oral Formulations of Levetiracetam in Healthy Male & Female Japanese Subjects
Brief Title: Human Pharmacology Study (Keppra Dry Syrup Bioequivalence Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: N01339
Record Dates: First submitted 2009-09-18; First posted 2009-09-28 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Levetiracetam; Healthy volunteers; Healthy Subjects
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment 1/Treatment 2 (Experimental)
  Interventions: Drug: Levetiracetam (Keppra)
- Treatment 2/Treatment 1 (Experimental)
  Interventions: Drug: Levetiracetam (Keppra)

INTERVENTIONS:
Drug: Levetiracetam (Keppra) — Test Drug :
  Levetiracetam dry syrup
  Reference Drug :
  500 mg oral tablets of Levetiracetam. Frequency: Single Dose
  Other Names: Keppra

SUMMARY:
To demonstrate the bioequivalence of a Levetiracetam dry syrup (50% (500mg/1000mg)) versus Levetiracetam 500 mg oral tablet, used as reference, after single dose administration in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent dated and signed by subject.
* Healthy male or female Japanese volunteer from the first generation, living outside of Japan for less than 10 years, age range 20 to 55 years inclusive.
* Body Mass Index (BMI) between 18.0 and 28.0 kg/m² inclusive.

Exclusion Criteria:

* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, neurological, psychiatric disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication.
* History of drug addiction or presence of drug addiction (positive drug screen) or excessive use of alcohol (weekly intake in excess of 21 units alcohol for male and 14 units alcohol for female; one unit alcohol equals one glass of beer or lager, a glass of wine or a measure of spirits), of psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
* Heavy caffeine drinker (drinking >5 cups of coffee or equivalent, approximately 500mg of caffeine per day).
* Smokers of more than 10 cigarettes per day or smokers not willing to abstain from smoking while in the clinic for each period.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum plasma concentration) of Levetiracetam. | 36 hours
AUC (0-t) (Area under the plasma concentration vs. time curve observed from time 0 h up to the last measurable data point) of Levetiracetam | 36 hours
AUC (Area under the curve extrapolated to infinity) of Levetiracetam | 36 hours

SECONDARY OUTCOMES:
tmax (time of maximum plasma concentration) of Levetiracetam | 36 hours
λz (Terminal elimination rate constant) of Levetiracetam | 36 hours
t1/2 (Terminal elimination half-life) of Levetiracetam | 36 hours
MRT (Mean Residence Time) of Levetiracetam | 36 hours
CL/F (Apparent total body clearance) of Levetiracetam | 36 hours
Vz/F (Apparent volume of distribution) of Levetiracetam | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- London, United Kingdom